CLINICAL TRIAL: NCT01204580
Title: ADIponectin and ADMA Level in Type-2 Diabetes Patients After 12 Weeks of Treatment With GlimepiRide And Metformin Fixed Dose Combination (Amaryl-M)
Brief Title: ADIponectin and Asymmetric Dimethylarginine (ADMA) Level in Type-2 Diabetes Patients After 12 Weeks of Treatment With GlimepiRide And Metformin Fixed Dose Combination
Acronym: DIAGRAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMET_L_04735; U1111-1116-8173 (Other: UTN)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

ARMS (1):
- Amaryl-M (Glimepiride + Metformin) (Experimental): Glimepiride 1 mg and metformin 250 mg are the active ingredients of Amaryl-M 1/250 mg film coated tablets.
  Starting dosage is 1 tablet per day, then dosage titration will be based on the result of patient FBG test.
  Interventions: Drug: GLIMEPIRIDE + METFORMIN

INTERVENTIONS:
Drug: GLIMEPIRIDE + METFORMIN — Pharmaceutical form: film coated tablet Route of administration: oral Dose regimen: 1 tablet of 1/250 mg per day
  Other Names: Amaryl-M

SUMMARY:
Primary Objective:

To evaluate the change in plasma levels of adiponectin and Asymmetric Dimethylarginine (ADMA) in type 2 diabetes patients after 12 weeks of treatment with Amaryl-M

Secondary Objectives:

1. To assess the role of Amaryl-M in the change of plasma levels of adiponectin and ADMA in type 2 diabetes patients after 8 weeks of therapy
2. To evaluate the brachial-ankle pulse wave velocity (baPWV) change after 8 and 12 weeks of therapy with Amaryl-M
3. To evaluate the efficacy of Amaryl-M in the improvement of patients glycemic level (Fasting blood glucose (FBG) and glycosylated hemoglobin (HbA1c))
4. To evaluate the change of Tumor Necrosis Factor - Alfa (TNF-Alfa) after 12 weeks of therapy with Amaryl-M
5. To evaluate the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) change after 12 weeks of therapy with Amaryl-M
6. To evaluate the HOMA-β change after 12 weeks of therapy with Amaryl-M
7. To evaluate the relationship between adiponectin and ADMA level with FBG or HbA1c level

DETAILED DESCRIPTION:
The clinical trial will consist of 2 weeks of selection followed by a 12 weeks (3 months) of treatment period.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus patients
* Patients with HbA1c >or= 7.0% and < 10.0%
* Patients not currently treated with any oral antidiabetic drugs (OADs)

Exclusion criteria:

* Participation in other investigational Clinical Trial
* Current temporary insulin treatment: gestational diabetes, pancreas cancer, surgery etc.
* Women who are pregnant and lactating
* Type 1 diabetes mellitus patients
* Treatment with antihypertensive Angiotensin-Converting Enzyme (ACE)-Inhibitors and/or Angiotensin II Receptor Blocker (ARB) or has just stopped treatment for less than two months
* Treatment with lipid lowering agent statins or has just stopped treatment for less than two months
* Known hypersensitive to any of the excipients of Amaryl-M, sulphonylureas, sulfonamides or biguanide
* Patients with active smoking or history of smoking cessation less than 2 months
* Patients with history of severe hepatic dysfunction
* Patients with serum creatinine >or= 1.5 mg/dL (male) and >or= 1.4 mg/dL (female)
* Patients with congestive heart failure requiring pharmacologic treatment
* Treatment with antifungal agent especially Miconazole

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adiponectin and Asymmetric Dimethylarginine (ADMA) plasma level changes | from baseline to end of Clinical Trial (12 weeks)

SECONDARY OUTCOMES:
Change in adiponectin and Asymmetric Dimethylarginine (ADMA) plasma levels | at week 8
Pulse Wave Velocity (PWV) change | at week 8 and week 12
Change in Fasting Blood Glucose (FBG) | At week 2, 4, 8 and 12
Change in glycosylated hemoglobin (HbA1c) | at week 12
Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) and Homeostatic Model Assessment (HOMA-β) | At week 12
Change of Tumor Necrosis Factor- Alfa (TNF-Alfa) | At week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Jakarta, Indonesia